CLINICAL TRIAL: NCT04322552
Title: A Single Arm, Open and Fixed Sequence Study to Investigate the Pharmacokinetic Effects of Apatinib Mesylate on Transporter Pgp Substrate Digoxin in Advanced Solid Tumor Subjects
Brief Title: A Pharmacokinetic Interaction Study Between Apatinib Mesylate and Transporter Pgp Substrate Digoxin in Advanced Solid Tumor Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-APTN-I-007
Record Dates: First submitted 2020-03-17; First posted 2020-03-26 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — apatinib; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treament (Experimental): In phase A, subjects receiving a single 0.25 mg of digoxin orally and wash-out for 5 days, then apatinib once daily will be conducted on D5 through D16 ； In addition, a single dose of 0.25 mg digoxin (in combination with apatinib) will be orally administered in fasting conditions on D12；
  Interventions: Drug: Apatinib Mesylate; Drug: Digoxin tablet

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib at a dosage of will be administered daily from on D5 through D16
Drug: Digoxin tablet — Digoxin at a dosage of 0.25mg will be administered at day 1 and day 12

SUMMARY:
Apatinib, an oral inhibitor of vascular endothelial growth factor receptor 2#VEGFR-2#, Induces Transporter Pgp function in vitro. This study in patients with advanced cancer evaluated the effect of Apatinib on Transporter Pgp function by comparing the pharmacokinetics of Transporter Pgp-specific probe drugs in the presence and absence of Apatinib. The probes used Substrate Digoxin.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of advanced solid tumors. 2. ECOG PS score: 0-1; 3. Expected survival ≥ 3 months; 4. Major organs must function normally, meeting the following criteria:

1. Hematology

   1. HB≥100 g/L;
   2. ANC≥1.5×109/L;
   3. PLT≥90×109/L;
2. Blood biochemistry:

   1. TBIL≤ 1.25×ULN;
   2. ALT and AST≤2.5×ULN;
   3. ALP≤2.5×ULN;
   4. Serum Cr ≤ 1.5 × ULN or endogenous CrCl ≥ 60 mL/min (Cockcroft-Gault formula);
   5. Albumin > 30 g/L;
   6. K+>3.0mmol/L; 5. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Primary liver cancer; gastric cancer;
2. Active brain metastasis (medically uncontrolled), carcinomatous meningitis, spinal cord compression;
3. Presence of clinically symptomatic third space fluid;
4. Uncontrolled hypertension (SBP ≥ 140 mmHg and/or DBP ≥ 90 mmHg despite optimal pharmacological treatment);
5. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) >2 NYHA 2 congestive heart failure; (2) left ventricular ejection fraction (LVEF) < 50% (3) heart rate <60 (4) Grade II or greater myocardial ischemia or myocardial infarction(5) QTc interval ≥ 450 ms in males and ≥ 470 ms in females;
6. Abnormal coagulation function;
7. Prior radiotherapy, systemic chemotherapy (< 6 weeks if chemotherapy including nitrosoureas or mitomycin), hormone therapy, surgery or target therapy within 4 weeks before the study drug administration, or any unresolved AEs > CTC-AE Grade 1;
8. History of psychotropic substance abuse, alcoholism or drug abuse;
9. Use of study drugs in other clinical trials within 4 weeks prior to the first dose；
10. Use of a potent CYP3A4 inhibitor or inducer within 2 weeks prior to the first dose;
11. Use of any prescription or over-the-counter medication, vitamin products or herbs within 2 weeks before taking the investigational drug;
12. Other factors that may lead to the termination of the participation in the study at the discretion of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of digoxin | through study completion, an average of 16 days
  Peak Plasma Concentration (Cmax) of digoxin
Pharmacokinetics parameter: AUC of digoxin | through study completion, an average of 16 days
  Area under the plasma concentration versus time curve (AUC) of digoxin

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax of digoxin | through study completion, an average of 16 days
  Time of maximum observed concentration (Tmax) of digoxin
Pharmacokinetics parameter: T1/2 of digoxin | through study completion, an average of 16 days
  Half time (T1/2) of digoxin
Pharmacokinetic parameters CL/F of digoxin | through study completion, an average of 16 days
  Total body clearance for extravascular administration (CL/F) of digoxin
Pharmacokinetics parameter: Vz/F of digoxin | through study completion, an average of 16 days
  Volume of distribution (Vz/F) of digoxin
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion, an average of 16 days
  An adverse event is any untoward medical occurrence in a patient or clinical study participant criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided